CLINICAL TRIAL: NCT00139659
Title: Efficacy and Safety of Inhaled Human Insulin (Exubera) Compared With Subcutaneous Human Insulin in the Therapy of Adult Subjects With Type 1 or Type 2 Diabetes Mellitus and Chronic Asthma: A One-Year, Multicenter, Randomized, Outpatient, Open-Label, Parallel-Group Comparative Trial
Brief Title: A One Year Clinical Trial Assessing the Usefulness and Safety of Inhaled Insulin in Diabetics With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171028
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Results first posted 2010-05-12 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2009-10

CONDITIONS: Asthma; Diabetes Mellitus
MeSH Terms: conditions — Asthma; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled Insulin (Experimental)
  Interventions: Drug: Inhaled Insulin
- Subcutaneous Insulin (Active Comparator)
  Interventions: Drug: Subcutaneous Insulin

INTERVENTIONS:
Drug: Inhaled Insulin — Inhaled insulin with dose adjusted according to premeal blood glucose plus oral antidiabetic agent(s) and/or either once or twice daily doses of either Ultralente or NPH insulin, or a single bedtime dose of insulin glargine.
  Arms: Inhaled Insulin
Drug: Subcutaneous Insulin — Subcutaneous short-acting insulin with dose adjusted according to premeal blood glucose plus oral antidiabetic agent(s) and/or either once or twice daily doses of either Ultralente or neutral protamine hagedorn (NPH) insulin, or a single bedtime dose of insulin glargine.
  Arms: Subcutaneous Insulin

SUMMARY:
A One Year Clinical Trial Assessing the Usefulness and Safety of Inhaled Insulin in Diabetics with Asthma

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus (Type 1 or Type 2) currently controlled with injected insulin
* Mild intermittent or mild to moderate persistent asthma

Exclusion Criteria:

* Poorly controlled, unstable or steroid-dependent asthma, insulin pump therapy, smoking

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2003-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (82):
- United States (67):
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Searcy, Arkansas
  - Pfizer Investigational Site, Berkeley, California
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Chiefland, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Honululu, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Normal, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Bossier City, Louisiana
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Waltham, Massachusetts
  - Pfizer Investigational Site, Brooklyn Center, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Butte, Montana
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, North Las Vegas, Nevada
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Lansdale, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Bartlett, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houstan, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Spokane, Washington
- Brazil (4):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Campinas, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
  - Pfizer Investigational Site, SP, São Paulo
- Canada (9):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Burlington, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Pfizer Investigational Site, San José, Provincia de San José, Costa Rica
- Pfizer Investigational Site, Neuss, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171028&StudyName=A%20One%20Year%20Clinical%20Trial%20Assessing%20the%20Usefulness%20and%20Safety%20of%20Inhaled%20Insulin%20in%20Diabetics%20with%20Asthma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 63 centers and participated in the study between 10 January 2003 and 22 October 2008.
Pre-assignment Details: 544 subjects were screened for the study. Prior to randomization subjects completed a 3-week run-in period during which all subjects received subcutaneous insulin. Of 288 subjects randomized, only 286 received randomized treatment; one subject assigned to inhaled insulin received subcutaneous insulin, and 1 subject DC'd prior to treatment.
Groups:
- Inhaled Insulin: Inhaled insulin (Exubera®) with dose adjusted according to premeal blood glucose plus basal insulin.
- Subcutaneous Insulin: Subcutaneous insulin with dose adjusted according to premeal blood glucose plus basal insulin.
Period: Overall Study
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Started | 146 (1 subject randomized was DC'd prior to receiving inhaled insulin but received subcutaneous insulin) | 141 (1 subject randomized DC'd before receiving subcutaneous insulin and is not included in # of subjects)
Completed | 106 | 123
Not Completed | 40 | 18
Not completed — Adverse Event | 12 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 7 | 3
Not completed — Reason not Specified | 6 | 3
Not completed — Withdrawal by Subject | 14 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Insulin | Subcutaneous Insulin | Total
Number analyzed (Participants) | 146 | 141 | 287
Age, Customized [Number; unit: participants]
  18-25 years | 12 | 8 | 20
  26-35 years | 18 | 13 | 31
  36-45 years | 23 | 25 | 48
  46-55 years | 33 | 41 | 74
  56-65 years | 40 | 37 | 77
  66-75 years | 20 | 17 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 91 | 188
  Male | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Change for Forced Expiratory Volume in 1 Second (FEV1)
Description: Annualized rates of change (slope throughout time from baseline to end of study[visit]) for forced expiratory volume in 1 second (FEV1) (liters per year [L/yr]) measured 30 minutes following the administration of albuterol.
Time Frame: Weeks -3, -2, -1, 1, 2, 3, 4, 6, 12, 18, 26, 39, and 52
Population: Primary analysis set (PAS): all subjects who were randomized, had no significant protocol violations, had baseline (BL) post-albuterol pulmonary function test (PFT) measurement, had at least 2 post-BL, post-albuterol PFT measurements with 1 measurement at least 6 months post-BL, and received study drug for at least 50% (154 days) of study duration.
Measure: Mean (Standard Error); unit: L/yr
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 117 | 127
L/yr | -0.070 (0.020) | -0.035 (0.019)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Treatment group difference (Exubera minus subcutaneous insulin): annualized rate of change over time. Longitudinal data analysis methods with random effects were used to model the pulmonary function test (PFT) measurements. Random effects included the intercept and slope with respect to time (visit); all remaining effects were fixed. The estimated rate of change over time for each treatment group was derived from this model; Test type: Superiority or Other; longitudinal data analysis model; Confidence interval of least squares (LS) mean difference (INH - SC) between annual rates of change for the two treatment groups; Mean Difference (Final Values) = -0.034, 90% CI [-0.080 to 0.011], Standard Error of Mean 0.028 — Primary analysis model includes terms of Treatment, Time, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on day of randomization

2. Secondary Outcome: Change From Baseline in Pre-Bronchodilator Forced Expiratory Volume in One Second (FEV1)
Description: Change from Baseline in Pre-Bronchodilator Forced Expiratory Volume in One Second (FEV1) at each visit. FEV1 was measured in liters (L) before the administration of albuterol. Change from baseline: mean FEV1 (L) at observation minus mean baseline value.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 6, Week 12, Week 18, Week 26, Week 39, Week 52, Week 52 Last Observation Carried Forward (LOCF)
Population: Full analysis set (FAS); LOCF: last observation carried forward.
Measure: Mean (Standard Error); unit: liters
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 141 | 139
liters
  Baseline (141, 139) | 2.435 (0.748) | 2.412 (0.727)
  Week 1 (123, 125) | -0.057 (0.142) | -0.035 (0.131)
  Week 2 (n=127, 117) | -0.065 (0.159) | -0.034 (0.150)
  Week 3 (n=130, 121) | -0.067 (0.185) | -0.044 (0.171)
  Week 4 (n=123, 130) | -0.076 (0.185) | -0.037 (0.181)
  Week 6 (n=130, 135) | -0.059 (0.211) | -0.034 (0.170)
  Week 12 (n=125, 130) | -0.067 (0.237) | -0.032 (0.193)
  Week 18 (n=125, 125) | -0.063 (0.218) | -0.042 (0.183)
  Week 26 (n=120, 129) | -0.058 (0.190) | -0.043 (0.195)
  Week 39 (n=108, 124) | -0.076 (0.195) | -0.044 (0.186)
  Week 52 (n=106, 112) | -0.136 (0.259) | -0.056 (0.230)
  Week 52 LOCF (n=141, 139) | -0.119 (0.259) | -0.058 (0.222)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 1; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.025, 90% CI [-0.065 to 0.015], Standard Error of Mean 0.024
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 2; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.034, 90% CI [-0.073 to 0.006], Standard Error of Mean 0.024
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 3; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.024, 90% CI [-0.063 to 0.016], Standard Error of Mean 0.024
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 4; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.035, 90% CI [-0.075 to 0.004], Standard Error of Mean 0.024
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 6; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.027, 90% CI [-0.067 to 0.012], Standard Error of Mean 0.024
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 12; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.033, 90% CI [-0.073 to 0.008], Standard Error of Mean 0.025
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 18; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.018, 90% CI [-0.059 to 0.023], Standard Error of Mean 0.025
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 26; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.010, 90% CI [-0.052 to 0.031], Standard Error of Mean 0.025
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 39; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.025, 90% CI [-0.068 to 0.017], Standard Error of Mean 0.026
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.073, 90% CI [-0.117 to -0.029], Standard Error of Mean 0.027
Statistical Analysis 11: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52 (LOCF); Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.061, 90% CI [-0.108 to -0.015], Standard Error of Mean 0.028

3. Secondary Outcome: Change From Baseline in Pre-Bronchodilator Carbon Monoxide Diffusing Capacity (DLco)
Description: Change From Baseline in Pre-Bronchodilator Carbon Monoxide Diffusing Capacity (DLco) measured in milliters/minutes/millimeters of mercury (mL/min/mmHg): change = DLco at observation minus DLco at Baseline.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 12, Week 18, Week 26, Week 39, Week 52, Week 52 Last Observation carried Forward (LOCF)
Population: Full analysis set (FAS); LOCF: last observation carried forward.
Measure: Mean (Standard Deviation); unit: ml/min/mmHg
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 141 | 139
ml/min/mmHg
  Baseline (n=141, 139) | 23.034 (5.921) | 22.911 (6.059)
  Week 1 (n=123, 125) | -0.749 (1.467) | -0.452 (1.220)
  Week 2 (n=126, 114) | -0.835 (1.353) | -0.456 (1.485)
  Week 3 (n=128, 119) | -0.855 (1.407) | -0.556 (1.452)
  Week 4 (n=122, 127) | -1.120 (1.609) | -0.648 (1.500)
  Week 6 (n=129, 135) | -1.169 (1.583) | -0.669 (1.441)
  Week 12 (n=124, 128) | -1.018 (1.842) | -0.725 (1.788)
  Week 18 (n=123, 125) | -0.906 (1.756) | -0.646 (1.748)
  Week 26 (n=117, 127) | -0.945 (1.683) | -0.561 (1.982)
  Week 39 (n=106, 125) | -0.821 (1.742) | -0.550 (1.805)
  Week 52 (n=105, 111) | -1.699 (2.157) | -0.911 (2.239)
  Week 52 LOCF (n=141, 139) | -1.557 (2.109) | -0.785 (2.141)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.327, 90% CI [-0.679 to 0.026], Standard Error of Mean 0.214
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.378, 90% CI [-0.729 to -0.027], Standard Error of Mean 0.213
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.346, 90% CI [-0.696 to 0.004], Standard Error of Mean 0.213
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.496, 90% CI [-0.847 to -0.145], Standard Error of Mean 0.213
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.610, 90% CI [-0.960 to -0.260], Standard Error of Mean 0.213
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.360, 90% CI [-0.721 to 0.001], Standard Error of Mean 0.219
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.291, 90% CI [-0.655 to 0.073], Standard Error of Mean 0.221
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.420, 90% CI [-0.788 to -0.052], Standard Error of Mean 0.224
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.337, 90% CI [-0.717 to 0.042], Standard Error of Mean 0.231
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.789, 90% CI [-1.181 to -0.397], Standard Error of Mean 0.238
Statistical Analysis 11: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.786, 90% CI [-1.178 to -0.393], Standard Error of Mean 0.238

4. Secondary Outcome: Change From Baseline in Pre-Insulin Forced Expiratory Volume in One Second (FEV1)
Description: Change from Baseline in Pre-Insulin Forced Expiratory Volume in one second (FEV1) measured in liters (L): change = FEV1 at observation minus FEV1 at Baseline.
Time Frame: Baseline, Week 9, Week 51, Week 51 Last Observation Carried Forward
Population: Full analysis set (FAS); LOCF: last observation carried forward.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 130 | 133
liters
  Baseline (n=130, 133) | 2.449 (0.775) | 2.403 (0.727)
  Week 9 (n=111, 108) | -0.038 (0.235) | -0.028 (0.163)
  Week 51 (n=103, 119) | -0.078 (0.227) | -0.017 (0.245)
  Week 51 LOCF (n=130, 133) | -0.068 (0.237) | -0.018 (0.237)

5. Secondary Outcome: Change From Baseline in Pre-Insulin Carbon Monoxide Diffusing Capacity (DLco)
Description: Change From Baseline in Pre-Insulin Carbon Monoxide Diffusing Capacity (DLco) measured in milliters/minutes/millimeters of mercury (mL/min/mmHg): change = DLco at observation minus DLco at Baseline.
Time Frame: Baseline, Week 9, Week 51, Week 51 Last Observation Carried Forward (LOCF)
Population: Full analysis set (FAS); LOCF: last observation carried forward.
Measure: Mean (Standard Deviation); unit: ml/min/mmHg
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 128 | 131
ml/min/mmHg
  Baseline (n=128, 131) | 22.836 (6.087) | 22.718 (6.128)
  Week 9 (n=109, 106) | -1.130 (1.663) | -0.663 (1.549)
  Week 51 (n=102, 116) | -1.156 (1.825) | -0.630 (2.023)
  Week 51 LOCF (n=128, 131) | -1.185 (1.804) | -0.533 (1.990)

6. Secondary Outcome: Change From Baseline in Post-bronchodilator Forced Vital Capacity (FVC)
Description: Change from baseline in Post-bronchodilator Forced Vital Capacity (FVC) measured in liters (L) 30 minutes following the administration of albuterol: change = FVC at observation minus FVC at Baseline.
Time Frame: as for outcome 3
Population: Full analysis set (FAS); LOCF: last observation carried forward.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 141 | 139
liters
  Baseline (n=141, 139) | 3.355 (0.963) | 3.341 (0.918)
  Week 1 (n=123, 125) | -0.068 (0.181) | -0.046 (0.134)
  Week 2 (n=126, 115) | -0.057 (0.190) | -0.053 (0.169)
  Week 3 (n=131, 119) | -0.078 (0.205) | -0.068 (0.174)
  Week 4 (n=121, 129) | -0.065 (0.193) | -0.051 (0.176)
  Week 6 (n=130, 135) | -0.092 (0.287) | -0.043 (0.173)
  Week 12 (n=125, 129) | -0.045 (0.222) | -0.056 (0.190)
  Week 18 (n=124, 125) | -0.053 (0.225) | -0.069 (0.179)
  Week 26 (n=120, 128) | -0.061 (0.215) | -0.052 (0.186)
  Week 39 (n=107, 124) | -0.080 (0.209) | -0.057 (0.213)
  Week 52 (n=106, 112) | -0.105 (0.288) | -0.088 (0.259)
  Week 52 LOCF (n=141, 139) | -0.097 (0.278) | -0.083 (0.247)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 1; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.021, 90% CI [-0.066 to 0.023], Standard Error of Mean 0.027
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 2; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.000, 90% CI [-0.044 to 0.044], Standard Error of Mean 0.027
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 3; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.012, 90% CI [-0.056 to 0.032], Standard Error of Mean 0.027
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 4; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.004, 90% CI [-0.048 to 0.041], Standard Error of Mean 0.027
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 6; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.045, 90% CI [-0.089 to -0.001], Standard Error of Mean 0.027
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 12; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.010, 90% CI [-0.035 to 0.056], Standard Error of Mean 0.028
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 18; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.018, 90% CI [-0.028 to 0.064], Standard Error of Mean 0.028
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 26; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.005, 90% CI [-0.051 to 0.041], Standard Error of Mean 0.028
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 39; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.022, 90% CI [-0.070 to 0.026], Standard Error of Mean 0.029
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.015, 90% CI [-0.064 to 0.034], Standard Error of Mean 0.030
Statistical Analysis 11: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52 (LOCF); Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.015, 90% CI [-0.067 to 0.037], Standard Error of Mean 0.031

7. Secondary Outcome: Bronchodilator Responsiveness as Determined by the Change in Forced Expiratory Volume in 1 Second (FEV1) Pre-albuterol and 30 Minutes Post-albuterol
Description: Responsiveness was the percent change from the forced expiratory volume in 1 second (FEV1) value before bronchodilator use to the FEV1 value 30 minutes after bronchodilator use, operationally defined as [(post-bronchodilator FEV1 minus pre-bronchodilator FEV1 divided by pre-bronchodilator FEV1] multiplied by 100.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 12, Week 18, Week 26, Week 39, Week 52
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: percent change in FEV1
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 141 | 139
percent change in FEV1
  Baseline (n=141, 139) | 5.487 (5.163) | 5.102 (6.416)
  Week 1 (n=123, 125) | -0.015 (5.452) | 0.347 (5.429)
  Week 2 (n=126, 115) | 0.683 (5.984) | 0.347 (6.354)
  Week 3 (n=130, 119) | -0.055 (6.082) | 0.823 (5.449)
  Week 4 (n=121, 129) | 0.056 (6.361) | 0.559 (5.733)
  Week 6 (n=130, 135) | -0.460 (5.480) | 0.504 (6.350)
  Week 12 (n=124, 129) | 0.721 (5.972) | -0.100 (6.783)
  Week 18 (n=124, 125) | -0.095 (5.909) | 0.154 (7.649)
  Week 26 (n=120, 128) | -0.186 (5.624) | 0.211 (5.080)
  Week 39 (n=107, 124) | -0.283 (5.368) | 0.133 (5.089)
  Week 52 (n=106, 112) | 0.640 (5.338) | -0.035 (6.156)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.632, 90% CI [-1.778 to 0.514], Standard Error of Mean 0.697
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.020, 90% CI [-1.079 to 1.120], Standard Error of Mean 0.668
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.582, 90% CI [-0.535 to 1.700], Standard Error of Mean 0.679
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.054, 90% CI [-1.184 to 1.077], Standard Error of Mean 0.687
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 6, analysis 5]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.535, 90% CI [-1.677 to 0.608], Standard Error of Mean 0.694
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.905, 90% CI [-2.014 to 0.203], Standard Error of Mean 0.674
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.212, 90% CI [-0.899 to 1.323], Standard Error of Mean 0.675
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 6, analysis 8]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.044, 90% CI [-1.080 to 1.169], Standard Error of Mean 0.683
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 6, analysis 9]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.240, 90% CI [-1.382 to 0.902], Standard Error of Mean 0.694
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.503, 90% CI [-1.673 to 0.668], Standard Error of Mean 0.711

8. Secondary Outcome: Percent Predicted and Percent Change From Baseline in Post-Bronchdilator Forced Expiratory Volume in One Second (FEV1)
Description: Percent predicted change from Baseline in post-bronchodilator forced expiratory volume in one second (FEV1) measured in liters (L): National Health and Nutrition Examination Survey (NHANES III) reference standard. Percent change from Baseline in post-bronchdilator FEV1 measured in liters (L): (observed value minus Baseline value) divided by Baseline value *100%.
Time Frame: as for outcome 3
Population: Full analysis set (FAS); LOCF: last observation carried forward.
Measure: Mean (Standard Deviation); unit: percentage of FEV1
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 141 | 139
percentage of FEV1
  Baseline (n=141, 139) | 83.698 (14.096) | 82.833 (15.219)
  Week 1: % of Predicted Value (n=123, 125) | 81.987 (14.441) | 82.878 (15.438)
  Week 2: % of Predicted Value (n=126, 115) | 81.655 (13.985) | 81.881 (15.017)
  Week 3: % of Predicted Value (n=131, 119) | 80.711 (13.854) | 82.036 (15.354)
  Week 4: % of Predicted Value (n=121, 129) | 81.093 (15.145) | 82.029 (14.914)
  Week 6: % of Predicted Value (n=130, 135) | 81.611 (14.553) | 82.016 (15.509)
  Week 12: % of Predicted Value (n=125, 129) | 82.145 (13.885) | 81.640 (14.673)
  Week 18: % of Predicted Value (n=124, 125) | 82.187 (14.405) | 81.723 (14.505)
  Week 26: % of Predicted Value (n=120, 128) | 82.941 (14.291) | 82.227 (14.305)
  Week 39: % of Predicted Value (n=107, 124) | 82.851 (14.447) | 81.847 (14.794)
  Week 52: % of Predicted Value (n=106, 112) | 80.869 (14.934) | 81.138 (14.461)
  Week 52 LOCF: % of Predicted Value (n=141, 139) | 80.136 (14.528) | 80.687 (14.671)
  Week 1: % Change from Baseline (n=123, 125) | -2.682 (5.780) | -1.238 (5.307)
  Week 2: % Change from Baseline (n=126, 115) | -2.355 (5.909) | -1.142 (5.273)
  Week 3: % Change from Baseline (n=131, 119) | -2.943 (7.583) | -1.057 (5.292)
  Week 4: % Change from Baseline (n=121, 129) | -3.063 (6.926) | -0.833 (6.172)
  Week 6: % Change from Baseline (n=130, 135) | -2.559 (8.725) | -0.957 (6.180)
  Week 12: % Change from Baseline (n=125, 129) | -1.975 (8.495) | -1.226 (7.603)
  Week 18: % Change from Baseline (n=124, 125) | -2.437 (8.713) | -1.247 (6.688)
  Week 26: % Change from Baseline (n=120, 128) | -2.006 (6.891) | -1.189 (8.013)
  Week 39: % Change from Baseline (n=107, 124) | -3.144 (7.507) | -1.466 (8.332)
  Week 52: % Change from Baseline (n=106, 112) | -4.777 (8.794) | -2.002 (10.040)
  Week 52 LOCF: % Change from Baseline (n=141, 139) | -4.129 (9.673) | -2.108 (9.652)

9. Secondary Outcome: Change From Baseline in Insulin Dose Responsiveness for Forced Expiratory Volume in One Second (FEV1) Measured 10 and 60 Minutes After the First Daily Dose of Insulin
Description: Change from Baseline in Insulin Dose Responsiveness for Forced Expiratory Volume in one second (FEV1) measured 10 and 60 minutes after the first daily dose of insulin. Insulin dose responsiveness = the difference between FEV1 value following a dose of insulin and FEV1 value before a dose of insulin, operationally defined as the post dose FEV1 value minus predose FEV1 value.
Time Frame: Baseline, Week 9, Week 51
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 124 | 131
liters
  Baseline: 10 minutes (n=124, 131) | -0.004 (0.085) | 0.003 (0.086)
  Week 9: 10 minutes (n=105, 106) | -0.008 (0.130) | 0.005 (0.111)
  Week 51: 10 minutes (n=96, 113) | 0.000 (0.113) | 0.013 (0.104)
  Baseline: 60 minutes (n=125, 131) | -0.004 (0.120) | 0.016 (0.130)
  Week 9: 60 minutes (n=105, 105) | 0.013 (0.113) | 0.028 (0.137)
  Week 51: 60 minutes (n=99, 112) | 0.029 (0.139) | 0.020 (0.123)

10. Secondary Outcome: Percent Predicted and Percent Change From Baseline in 10 Minute and 60 Minute Post-Insulin Forced Expiratory Volume in One Second (FEV1)
Description: Percent predicted change from Baseline in 10 Minute and 60 Minute post-insulin forced expiratory volume in one second (FEV1) measured in liters (L): National Health and Nutrition Examination Survey (NHANES III) reference standard. Percent change from Baseline in FEV1 measured in liters (L) 10 and 60 Minutes post-insulin. Percent change = (value at observation minus Baseline value) divided by Baseline value *100%.
Time Frame: Baseline, Week 9, Week 51, Week 51 Last Observation Carried Forward (LOCF)
Population: Full analysis set (FAS); LOCF: last observation carried forward.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 124 | 131
percent
  Baseline: 10 minutes (n=124, 131) | 94.402 (6.532) | 94.391 (6.168)
  Week 9: 10 min.; % of Predicted Value (n=105, 106) | 92.698 (9.187) | 94.190 (7.190)
  Week 9: 10 min;% Change from Baseline (n=105, 106) | -1.864 (9.684) | -0.456 (8.638)
  Week 51: 10 min.;% of Predicted Value (n=96, 113) | 91.668 (8.223) | 93.717 (9.305)
  Week 51:10 min;% Change from Baseline (n=96, 113) | -2.760 (8.789) | 0.228 (13.653)
  Week 51 LOCF:10 min;% Predicted Value (n=124, 131) | 91.196 (8.366) | 93.882 (9.013)
  Week 51 LOCF:10 min;% Change from BL (n=124, 131) | -3.176 (8.825) | -0.029 (12.946)
  Baseline: 60 minutes (n=125, 131) | 94.284 (6.548) | 94.688 (5.260)
  Week 9: 60 min.; % of Predicted Value (n=105, 105) | 93.586 (8.219) | 94.950 (7.526)
  Week 9: 60 min;% Change from Baseline (n=105, 105) | -0.450 (9.464) | -0.031 (7.497)
  Week 51: 60 min.; % of Predicted Value (n=99, 112) | 92.302 (7.949) | 94.084 (9.069)
  Week 51:60 min.;% Change from Baseline (n=99, 112) | -1.699 (9.015) | -0.247 (10.349)
  Week 51 LOCF:60 min;% Predicted Value (n=125, 131) | 92.418 (8.544) | 94.300 (8.823)
  Week 51 LOCF:60 min;% Change from BL (n=125, 131) | -1.714 (9.512) | -0.222 (9.816)

11. Secondary Outcome: Change From Baseline in Insulin Dose Responsiveness for Carbon Monoxide Diffusing Capacity (DLco) Measured 10 and 60 Minutes After the First Daily Dose of Insulin
Description: Carbon Monoxide Diffusing Capacity (DLco) dose responsivness 10 and 60 minutes after insulin. DLco dose-responsiveness to insulin was defined as the difference between the DLco value following a dose of insulin and DLco value before a dose of insulin, operationally defined as the post-dose DLco value minus pre-dose DLco value.
Time Frame: Baseline, Week 9, Week 51
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: ml/min/mmHg
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 122 | 129
ml/min/mmHg
  Baseline: 10 minutes (n=122, 129) | -0.163 (0.992) | -0.184 (0.985)
  Week 9: 10 minutes (n=102, 104) | -0.241 (1.390) | -0.131 (1.006)
  Week 51: 10 minutes (n=95, 109) | -0.139 (0.893) | -0.171 (0.820)
  Baseline: 60 minutes (n=135, 133) | -0.446 (1.115) | -0.451 (1.258)
  Week 9: 60 minutes (n=104, 108) | -0.338 (1.416) | -0.159 (1.126)
  Week 51: 60 minutes (n=101, 110) | -0.216 (1.458) | -0.383 (1.030)

12. Secondary Outcome: Methacholine Challenge
Description: Methacholine Challange: performed on a subset of subjects using the 5-breath dosimeter method. Subjects were challenged with ascending doses of nebulized methacholine; dosing schedule: 0.03, 0.06, 0.12, 0.25, 0.5, 1.0, 2.0, 4.0, 8.0, 16.0, 32.0 milligrams per milliliter (mg/ml) administered in 5-minute intervals. Forced expiratory volume in 1 second (FEV1) was measured 1-3 minutes after each inhalation of methacholine solution. Testing continued until highest FEV1 decreased by ≥20% from the challenge (post-diluent) reference, or until completion all doses.
Time Frame: 1 to 2 days following Weeks -3 and -1 visits, and at Week 11, Week 50, and Week 52 (+5)
Population: There were no methacholine challenges performed in subjects using inhaled insulin due to protocol-defined exclusion criteria for methacholine challenge testing, and methacholine provocative concentration [of methacholine] causing a 20% fall in FEV1 (PC20) data were not analyzed.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Mean Weekly Morning and Evening Peak Expiratory Flow Rate (PEFR) and Forced Expiratory Volume in 1 Second (FEV1)
Description: Subjects measured peak expiratory flow rate (PEFR) and forced expiratory volume in 1 second (FEV1) twice daily and entered the results in an electronic diary. Daily data were used to calculate the mean PEFR and FEV1 for each week (observed weekly mean and change from baseline in weekly mean). For each subject, the mean weekly morning (and evening) PEFR and FEV1 was defined as the sum of the daily morning (and evening) PEFR (and FEV1) measurements during the week divided by the number of non-missing PEFR (and FEV1) measurements during the week.
Time Frame: Week -3 through Week 52
Population: Mean weekly morning and evening peak expiratory flow rate (PEFR) and forced expiratory volume in 1 second (FEV1) were not presented due to lack of resource resulting from scaling down of Exubera® (inhaled insulin) development.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Mean Weekly Number of Puffs of Albuterol Used (Rescue Medication)
Description: All subjects used an electronic symptom diary to record their daily use of short-acting bronchodilators. Subjects recorded the sum of their short-acting bronchodilator use (puffs of albuterol) daily, immediately upon arising, and again in the evening or before bed.
Time Frame: Daily: Baseline to end of study
Population: Mean weekly number of puffs of albuterol was not presented due to lack of resource resulting from scaling down of Exubera® (inhaled insulin) development.
Measure: Mean (Standard Deviation); unit: number of puffs
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Subjects With Step-up and Step-down Changes in Classification of Asthma Severity by Medication Usage
Description: All asthma medication changes during the study were classified as step-up or step-down according to treatment guidelines. Step 1: Intermittant Asthma; Step 2: Mild Persistent Asthma; Step 3: Moderate Persistent Asthma; Step 4: Severe Persistent Asthma. The number of subjects in each step classification of asthma severity were provided at each assessment timepoint for each treatment group, with a shift table indicating the number of subjects moving from each step classification at each timepoint.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 6, Week 9, Week 12, Week 18, Week 26, Week 39, Week 52, Week 54, Week 58
Population: Data for the number of step-up and step-down changes in classification of asthma severity by medication usage were not tabulated or analyzed as accurate dose information data for all concomitant medications were not available due to inconsistencies in the way concomitant medication data were collected.
Measure: Number; unit: subjects
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Step Classification of Asthma Severity by Medication Usage
Description: Step classification of asthma severity by medication usage. Subjects were classified at each visit according to the medication used on the day of the particular time-point; Step 1: intermittent asthma, Step 2: mild persistent asthma, Step 3: moderate persistent asthma, Step 4: severe persistent asthma. The number (%) of subjects in each step classification were provided at each assessment timepoint with a shift table indicating the number (%) of subjects moving from each step classification at each time-point.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 6, Week 9, Week 12, Week 18, Week 26, Week 39, Week 52, Week 54, Week 58
Population: Data for step classification of asthma severity by medication usage were not tabulated or analyzed as accurate dose information data for all concomitant medications were not available due to inconsistencies in the way concomitant medication data were collected.
Measure: Number; unit: subjects
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Mean Weekly Asthma Symptom Scores
Description: Mean weekly asthma symptom scores: subjects recorded their asthma symptom scores in an electronic symptom diary twice daily throughout the study, immediately upon awakening (5-10 AM) and in the evening or at bedtime (7-12 PM). Questions included extent of albuterol use, symptoms of wheezing, coughing, activity limitations and sleep; scale 0 (none/fine) to 3 (severe/ continuous/bad night).
Time Frame: Baseline through end of study
Population: Data for mean weekly asthma symptom scores were not presented due to lack of resource resulting from scaling down of Exubera® (inhaled insulin) development.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Incidence of Non-severe Asthma Exacerbations
Description: Non-severe asthma exacerbation = one of the following: any home monitored morning (4:45 am - 10:15 am) forced expiratory volume in 1 second (FEV1) <80% of the morning baseline for 2 or more consecutive days; or home monitored FEV1 <60% of Baseline at any time. Percent of Baseline = 100*(daily FEV1)/Baseline weekly FEV1. Subject-months=elapsed number of months a subject was in the study in each time interval. Crude event rate = total events divided by subject-months.
Time Frame: 0 to 1 week to > 12 months
Population: FAS; review of source data for this endpoint showed excessive data variability for home-monitored FEV1 with outliers ranging from 0.01 to >100, and many subjects with random peaks and dips of 100% or more of their baseline. It is unlikely that the protocol definition is robust enough to provide real information about exacerbation frequencies.
Measure: Number; unit: events/subject-months
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 141 | 139
events/subject-months
  0 to 1 Week (n=141, 139) | 0.43 | 0.41
  >1 to 2 Weeks (n=141, 139) | 0.28 | 0.38
  >2 to 3 Weeks (n=141, 139) | 0.22 | 0.31
  >3 to 4 Weeks (n=141, 139) | 0.37 | 0.41
  >4 to 6 Weeks (n=141, 139) | 0.52 | 0.36
  >6 to 9 Weeks (n=138, 139) | 0.53 | 0.51
  >9 to 12 Weeks (n=134, 138) | 0.35 | 0.46
  >3 Months (n=133, 137) | 0.40 | 0.40
  >6 to 9 Months (n=121, 133) | 0.30 | 0.49
  >9 to 12 Months (n=114, 131) | 0.27 | 0.43
  >12 Months (n=67, 81) | 0.34 | 0.21
  Overall (n=141, 139) | 0.35 | 0.43

19. Secondary Outcome: Incidence of Severe Asthma Exacerbations
Description: Severe asthma exacerbation was defined as one of the following: subject received oral (systemic) corticosteriods for the treatment of asthma; or subject had an unscheduled visit to a physician, emergency room, or hospital for the treatment of asthma. Subject-months=elapsed number of months a subject was in the study in each time interval. Crude event rate = total events divided by subject-months * 100.
Time Frame: 0 to 1 Week to > 12 Months
Population: Full analysis set (FAS); due to inconsistencies in data entry for systemic steroids, the protocol definition for severe asthma exacerbations, which was based on systemic corticosteroid use for asthma, could not be accurately assessed. Due the small number of events the incidence of severe asthma exacerbations was assessed per 100 months.
Measure: Number; unit: events/subject months*100
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 141 | 139
events/subject months*100
  0 to 1 Week (n=141, 139) | 0.00 | 0.00
  >1 to 2 Weeks (n=141, 139) | 0.00 | 3.13
  >2 to 3 Weeks (n=141, 139) | 0.00 | 9.39
  >3 to 4 Weeks (n=141, 139) | 3.08 | 0.00
  >4 to 6 Weeks (n=141, 139) | 4.63 | 1.56
  >6 to 9 Weeks (n=138, 139) | 1.06 | 0.00
  >9 to 12 Weeks (n=134, 138) | 1.09 | 0.00
  >3 Months (n=133, 137) | 1.20 | 2.27
  >6 to 9 Months (n=121, 133) | 1.43 | 1.01
  >9 to 12 Months (n=114, 131) | 1.53 | 1.33
  >12 Months (n=67, 81) | 3.39 | 0.00
  Overall (n=141, 139) | 1.46 | 1.47

20. Secondary Outcome: Number of Systemic Corticosteroid Rescues
Description: Number of subjects who used a systemic corticosteroid at any time during the study, and the total number of systemic corticosteroid rescues. New rescue event = >=2 consecutive days between the end of one event and the start of another event.
Time Frame: Baseline through Week 52
Population: Full analysis set (FAS); number of subjects with systemic corticosteroid rescues = inhaled insulin: 12, and subcutaneous insulin: 14. Due to inconsistencies in data entry, the numbers of systemic corticosteroid rescues were not considered entirely accurate.
Measure: Number; unit: systemic corticosteriod rescues
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 141 | 139
systemic corticosteriod rescues | 14 | 16

21. Primary Outcome: Annualized Rate of Change for Hemoglobin-adjusted Carbon Monoxide Diffusion Capacity (DLco)
Description: Annualized rates of change (slope throughout time from baseline to end of study[visit]) for hemoglobin-adjusted carbon monoxide diffusion capacity (DLco)in milliliters per minute/millimeters of mercury/year (ml/min/mmHg/yr) measured 30 minutes following the administration of albuterol.
Time Frame: Weeks -3, -2, -1, 1, 2, 3, 4, 6, 12, 18, 26, 39, and 52
Population: Primary analysis set (PAS).
Measure: Mean (Standard Error); unit: ml/min/mmHg/yr
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 117 | 127
ml/min/mmHg/yr | -0.776 (0.152) | -0.273 (0.153)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Longitudinal data analysis model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.503, 90% CI [-0.858 to -0.148], Standard Error of Mean 0.216 — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Asthma Control as Measured by the Asthma Control Questionnaire©
Description: Asthma Control Questionnaire©: 6 self-administered questions that assess asthma control over the past week covering nocturnal waking, morning symptoms, activity limitations, shortness of breath, wheezing, and short-acting bronchodilator use; 7-point ordinal rating scale from 0 (good control) to 6 (poor control). A seventh question was completed by a health professional on forced expiratory volume in 1 second (FEV1) % predicted using a one-week recall period; scale: 0 (>95% predicted) to 6 (<50% predicted). Overall score = mean of questions 1 - 7.
Time Frame: Baseline, Weeks 4, 12, 26, 39, 52
Population: FAS; abbreviations: Eval = evaluations, BL = Baseline.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 138 | 138
scores on scale
  Baseline: Subject Evaluation (n=138, 138) | 1.04 (0.78) | 1.21 (0.91)
  Baseline: Clinical Evaluation (n=138, 138) | 2.50 (1.50) | 2.54 (1.70)
  Baseline: Overall Evaluation (n=138, 138) | 1.25 (0.74) | 1.40 (0.86)
  Week 4: Subject Evaluation (n=123, 121) | 1.08 (0.81) | 1.15 (0.89)
  Week 4: Clinical Evaluation (n=123, 121) | 2.68 (1.52) | 2.65 (1.61)
  Week 4: Overall Evaluation (n=123, 121) | 1.31 (0.78) | 1.36 (0.81)
  Week 12: Subject Evaluation (n=129, 134) | 1.04 (0.83) | 1.17 (0.91)
  Week 12: Clinical Evaluation (n=129, 134) | 2.55 (1.50) | 2.61 (1.48)
  Week 12: Overall Evaluation (n=129, 134) | 1.25 (0.77) | 1.37 (0.83)
  Week 26: Subject Evaluation (n=121, 131) | 1.06 (0.80) | 1.07 (0.91)
  Week 26: Clinical Evaluation (n=121, 131) | 2.48 (1.43) | 2.61 (1.57)
  Week 26: Overall Evaluation (n=121, 131) | 1.27 (0.74) | 1.29 (0.85)
  Week 39: Subject Evaluation (n=110, 125) | 0.94 (0.76) | 1.00 (0.85)
  Week 39: Clinical Evaluation (n=110, 125) | 2.54 (1.43) | 2.63 (1.52)
  Week 39: Overall Evaluation (n=110, 125) | 1.17 (0.71) | 1.23 (0.81)
  Week 52: Subject Evaluation (n=107, 120) | 1.08 (1.07) | 0.98 (0.84)
  Week 52: Clinical Evaluation (n=107, 120) | 2.77 (1.54) | 2.64 (1.56)
  Week 52: Overall Evaluation (n=107, 120) | 1.32 (0.99) | 1.21 (0.80)
  Week 4: Subject Eval: Change from BL (n=122, 120) | 0.02 (0.59) | -0.07 (0.59)
  Week 4: Clinical Eval: Change from BL (n=122, 120) | 0.17 (0.85) | 0.14 (0.85)
  Week 4: Overall Eval: Change from BL (n=122, 120) | 0.04 (0.55) | -0.04 (0.53)
  Week 12: Subject Eval: Change from BL (n=129, 134) | -0.02 (0.66) | -0.04 (0.72)
  Week 12 Clinical Eval: Change from BL (n=129, 134) | 0.12 (0.94) | 0.09 (0.91)
  Week 12: Overall Eval: Change from BL (n=129, 134) | 0.00 (0.59) | -0.02 (0.62)
  Week 26: Subject Eval: Change from BL (n=121, 130) | 0.05 (0.77) | -0.12 (0.82)
  Week 26 Clinical Eval: Change from BL (n=121, 130) | 0.09 (0.78) | 0.09 (1.00)
  Week 26: Overall Eval: Change from BL (n=121, 130) | 0.05 (0.68) | -0.09 (0.73)
  Week 39: Subject Eval: Change from BL (n=110, 124) | -0.09 (0.65) | -0.19 (0.77)
  Week 39 Clinical Eval: Change from BL (n=110, 124) | 0.14 (1.05) | 0.11 (0.94)
  Week 39: Overall Eval: Change from BL (n=110, 124) | -0.06 (0.58) | -0.15 (0.68)
  Week 52: Subject Eval: Change from BL (n=106, 119) | 0.06 (0.88) | -0.19 (0.86)
  Week 52 Clinical Eval: Change from BL (n=106, 119) | 0.38 (0.87) | 0.10 (1.20)
  Week 52: Overall Eval: Change from BL (n=106, 119) | 0.11 (0.77) | -0.15 (0.77)

23. Secondary Outcome: Baseline Dyspnea Index (BDI)
Description: Total score = the sum of the numeric grades from the three dyspnea index questions. Functional Impairment rating scale: Grade 4 (no impairment) to Grade 0 (very severe impairment); Magnitude of Task rating scale: Grade 4 (extraordinary) to Grade 0 (no task); and Magnitude of Effort rating scale: Grade 4 (extraordinary) to grade 0 (no effort).
Time Frame: run-in period
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 139 | 138
scores on scale
  Functional Impairment | 3.37 (0.80) | 3.36 (0.87)
  Magnitude of Task | 2.29 (1.19) | 2.29 (1.25)
  Magnitude of Effort | 2.49 (1.39) | 2.34 (1.49)
  Total Score | 8.15 (2.98) | 7.97 (2.99)

24. Secondary Outcome: Transition Dyspnea Index (TDI): Change in Total Score
Description: Transition Dyspnea Index total score = sum of the numeric grades from the three dyspnea index questions: Change in Functional Impairment, Change in Magnitude of Task, and Change in Magnitude of Effort. Rating scale: -3 (major deterioration), -2 (moderate deterioration), -1 (minor deterioration, 0 (no change), +1 (minor improvement), +2 (moderate improvement), +3 (major improvement).
Time Frame: Week 4, Week 12, Week 26, Week 39, Week 52
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 131 | 135
scores on scale
  Week 4 (n=121, 122) | 0.36 (1.93) | 0.50 (1.92)
  Week 12 (n=131, 135) | 0.51 (1.76) | 0.47 (1.68)
  Week 26 (n=124, 131) | 0.14 (1.75) | 0.13 (1.55)
  Week 39 (n=112, 127) | 0.26 (1.56) | 0.29 (1.61)
  Week 52 (n=105, 121) | 0.13 (1.65) | 0.67 (2.01)

25. Secondary Outcome: Glycosylated Hemoglobin (HbA1c)
Description: Glycosylated Hemoglobin (HbA1c): observed mean values at Baseline and each observation, and change from Baseline. Change from Baseline = mean HbA1c at observation minus mean HbA1c at Baseline.
Time Frame: Baseline, Week 6, Week 12, Week 26, Week 39, Week 52, Week 52 Last Observation Carried Forward (LOCF)
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 135 | 135
percent
  Baseline (n=135, 135) | 7.62 (1.12) | 7.43 (1.08)
  Week 6: Observed Value (n=127, 126) | 7.22 (1.00) | 6.97 (0.90)
  Week 6: Change from Baseline (n=127, 126) | -0.38 (0.65) | -0.43 (0.49)
  Week 12: Observed Value (n=122, 127) | 7.28 (1.12) | 6.98 (0.97)
  Week 12: Change from Baseline (n=122, 127) | -0.32 (0.98) | -0.48 (0.69)
  Week 26: Observed Value (n=118, 120) | 7.38 (1.24) | 7.19 (1.18)
  Week 26: Change from Baseline (n=118, 120) | -0.12 (1.07) | -0.25 (0.93)
  Week 39: Observed Value (n=108, 123) | 7.44 (1.31) | 7.20 (1.16)
  Week 39: Change from Baseline (n=108, 123) | -0.08 (1.10) | -0.21 (0.91)
  Week 52: Observed Value (n=101, 118) | 7.51 (1.35) | 7.35 (1.28)
  Week 52: Change from Baseline (n=101, 118) | 0.00 (1.05) | -0.05 (1.01)
  Week 52 (LOCF): Observed Value (n=135, 135) | 7.58 (1.35) | 7.40 (1.36)
  Week 52 (LOCF): Change from Baseline (n=135, 135) | -0.04 (1.07) | -0.03 (1.04)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 6; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of treatment, Week, Baseline HbA1c, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 90% CI [-0.06 to 0.28], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 12; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of treatment, Week, Baseline HbA1c, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.21, 90% CI [0.04 to 0.38], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 26; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of treatment, Week, Baseline HbA1c, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.17, 90% CI [-0.01 to 0.34], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 39; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of treatment, Week, Baseline HbA1c, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.14, 90% CI [-0.03 to 0.32], Standard Error of Mean 0.11
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52; Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of treatment, Week, Baseline HbA1c, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.06, 90% CI [-0.12 to 0.24], Standard Error of Mean 0.11
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52 (LOCF); Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of treatment, Week, Baseline HbA1c, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 90% CI [-0.19 to 0.22], Standard Error of Mean 0.12

26. Secondary Outcome: Fasting Plasma Glucose
Description: Fasting plasma glucose (milligrams per deciliter [mg/dL]) at Baseline, and change from Baseline. Change from baseline: mean of value of fasting plasma glucose in mg/dL at observation minus baseline value.
Time Frame: Baseline, Week 6, Week 12, Week 26, Week 39, Week 52, Week 52 Last Observation Carried Forward (LOCF)
Population: Primary analysis set (PAS); Last Observation Carried Forward: if the end of study value was missing the last available observation for that subject was used..
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 112 | 123
mg/dL
  Baseline (n=112, 123) | 149.22 (49.92) | 149.03 (58.33)
  Week 6: Observed Value (n=103, 112) | 143.02 (68.92) | 136.54 (57.98)
  Week 6: Change from Baseline (n=103, 112) | -3.34 (68.47) | -15.19 (67.16)
  Week 12: Observed Value (n=106, 113) | 136.32 (63.00) | 144.47 (61.22)
  Week 12: Change from Baseline (n=106, 113) | -12.16 (65.62) | -5.40 (67.71)
  Week 26: Observed Value (n=102, 114) | 139.05 (64.63) | 143.54 (52.09)
  Week 26: Change from Baseline (n=102, 114) | -11.86 (76.07) | -4.63 (65.10)
  Week 39: Observed Value (n=102, 115) | 143.64 (63.89) | 142.91 (66.26)
  Week 39: Change from Baseline (n=102, 115) | -5.67 (67.65) | -7.47 (65.55)
  Week 52: Observed Value (n=98, 115) | 146.32 (66.04) | 145.43 (59.35)
  Week 52: Change from Baseline (n=98, 115) | -3.86 (60.61) | -2.53 (63.23)
  Week 52 LOCF: Observed Value (n=112, 123) | 148.28 (71.07) | 144.96 (58.80)
  Week 52 LOCF: Change from Baseline (n=112, 123) | -0.95 (72.53) | -4.07 (62.75)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 6; Analysis of change from Baseline in fasting plasma glucose: Inhaled Insulin - Subcutaneouas Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline, Fasting Plasma Glucose, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Confidence interval for the LS mean of that particular treatment; Mean Difference (Final Values) = 10.615, 90% CI [-2.351 to 23.581], Standard Error of Mean 7.874
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 12; Analysis of change from Baseline in fasting plasma glucose: Inhaled Insulin - Subcutaneouas Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline, Fasting Plasma Glucose, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -6.942, 90% CI [-19.79 to 5.909], Standard Error of Mean 7.804
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 26; Analysis of change from Baseline in fasting plasma glucose: Inhaled Insulin - Subcutaneouas Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline, Fasting Plasma Glucose, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -4.622, 90% CI [-17.63 to 8.382], Standard Error of Mean 7.897
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 39; Analysis of change from Baseline in fasting plasma glucose: Inhaled Insulin - Subcutaneouas Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline, Fasting Plasma Glucose, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.828, 90% CI [-11.16 to 14.817], Standard Error of Mean 7.888
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52; Analysis of change from Baseline in fasting plasma glucose: Inhaled Insulin - Subcutaneouas Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline, Fasting Plasma Glucose, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.149, 90% CI [-12.01 to 14.307], Standard Error of Mean 7.991
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52 (LOCF); Analysis of change from Baseline in fasting plasma glucose: Inhaled Insulin - Subcutaneouas Insulin. Adjusted (Primary Analysis Model): includes terms of Treatment, Week, Baseline, Fasting Plasma Glucose, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 4.247, 90% CI [-8.664 to 17.157], Standard Error of Mean 7.816

27. Secondary Outcome: Body Weight: Mean Baseline and Change From Baseline
Description: Body weight: mean Baseline and change from Baseline in kilograms (kg). Change from baseline = mean body weight in kilograms (kg) at observation minus baseline value.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 9, Week 11, Week 12, Week 18, Wek 26, Week 39, Week 50, Week 51, Week 52, Week 52 Last Observation Carried Forward (LOCF)
Population: Primary analysis set (PAS)
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 113 | 124
kilograms
  Baseline (n=113, 124) | 87.41 (21.04) | 87.13 (17.58)
  Week 1: Change from Baseline (n=102, 113) | -0.02 (1.45) | 1.00 (7.63)
  Week 2: Change from Baseline (n=104, 105) | 0.12 (1.31) | 0.57 (1.50)
  Week 3: Change from Baseline (n=103, 113) | 0.18 (1.64) | 0.34 (1.55)
  Week 4: Change from Baseline (n=101, 119) | 0.31 (1.74) | 0.44 (1.70)
  Week 6: Change from Baseline (n=106, 122) | 0.13 (1.93) | 0.68 (1.88)
  Week 9: Change from Baseline (n=101, 104) | 0.14 (2.31) | 0.91 (2.33)
  Week 11: Change from Baseline (n=14, 17) | 0.71 (1.77) | 0.69 (2.00)
  Week 12: Change from Baseline (n=106, 118) | 0.01 (2.96) | 0.84 (2.83)
  Week 18: Change from Baseline (n=110, 116) | 0.35 (3.04) | 1.27 (3.46)
  Week 26: Change from Baseline (n=111, 121) | 0.72 (3.52) | 1.29 (3.32)
  Week 39: Change from Baseline (n=107, 121) | 0.77 (4.33) | 1.33 (3.70)
  Week 50: Change from Baseline (n=19, 13) | 0.04 (3.67) | 1.98 (3.90)
  Week 51: Change from Baseline (n=49, 60) | 0.24 (3.75) | 0.63 (4.38)
  Week 52: Change from Baseline (n=90, 109) | 1.34 (3.98) | 1.26 (4.08)
  Week 52 LOCF: Change from Baseline (n=113, 124) | 1.13 (3.95) | 1.44 (4.13)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 1; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.080, 90% CI [-1.829 to -0.331], Standard Error of Mean 0.455
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 2; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.475, 90% CI [-1.233 to 0.284], Standard Error of Mean 0.461
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 3; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.185, 90% CI [-0.931 to 0.562], Standard Error of Mean 0.454
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 4; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.189, 90% CI [-0.929 to 0.550], Standard Error of Mean 0.449
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 6; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.558, 90% CI [-1.294 to 0.178], Standard Error of Mean 0.447
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 9; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.748, 90% CI [-1.517 to 0.022], Standard Error of Mean 0.467
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 11; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.053, 90% CI [-2.510 to 0.405], Standard Error of Mean 0.886
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 12; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.891, 90% CI [-1.634 to -0.149], Standard Error of Mean 0.451
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 18; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.980, 90% CI [-1.725 to -0.234], Standard Error of Mean 0.453
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 26; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.663, 90% CI [-1.400 to 0.075], Standard Error of Mean 0.448
Statistical Analysis 11: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 39; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.537, 90% CI [-1.279 to 0.205], Standard Error of Mean 0.451
Statistical Analysis 12: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 50; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.322, 90% CI [-3.012 to 0.369], Standard Error of Mean 1.027
Statistical Analysis 13: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 51; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.063, 90% CI [-0.847 to 0.972], Standard Error of Mean 0.552
Statistical Analysis 14: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52; adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.193, 90% CI [-0.964 to 0.579], Standard Error of Mean 0.469
Statistical Analysis 15: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52 (LOCF); adjusted mean difference between inhaled insulin and subcutaneous insulin groups. Primary analysis model includes terms of Treatment, Week, Baseline Body Weight, Center, and Type of Diabetes; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.430, 90% CI [-1.298 to 0.438], Standard Error of Mean 0.526

28. Secondary Outcome: Total Daily Long-Acting Insulin Dose (Unadjusted for Body Weight)
Description: Total Daily Long-Acting Insulin Dose Unadjusted for Body Weight: long-acting insulin included Insulin NPH, Ultralente, and Insulin Glargine for both groups.
  Inhaled Insulin reported in mg. Subcutaneous Insulin reported in units.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 9, Week 12, Week 18, Week 26, Week 39, Week 52
Population: Primary analysis set (PAS)
Measure: Mean (Standard Deviation); unit: mg, units
Groups:
- Inhaled Insulin (mg): Inhaled insulin (Exubera®) with dose adjusted according to premeal blood glucose plus basal insulin.
- Subcutaneous Insulin (Units): Subcutaneous insulin with dose adjusted according to premeal blood glucose plus basal insulin.
Arm/Group | Inhaled Insulin (mg) | Subcutaneous Insulin (Units)
Number analyzed (Participants) | 111 | 122
mg, units
  Baseline (n=105, 121) | 41.70 (24.61) | 45.50 (27.54)
  Week 1 (n=104, 117) | 41.75 (25.75) | 45.46 (28.69)
  Week 2 (n=106, 111) | 43.48 (26.76) | 47.19 (28.08)
  Week 3 (n=104, 117) | 43.75 (27.32) | 47.61 (29.06)
  Week 4 (n=104, 120) | 44.70 (28.06) | 48.54 (29.91)
  Week 6 (n=106, 122) | 45.89 (29.31) | 48.59 (30.68)
  Week 9 (n=104, 109) | 46.01 (30.57) | 47.68 (29.16)
  Week 12 (n=110, 122) | 46.05 (30.82) | 49.04 (30.99)
  Week 18 (n=110, 120) | 47.15 (32.34) | 49.94 (30.95)
  Week 26 (n=111, 122) | 47.65 (33.87) | 49.98 (31.32)
  Week 39 (n=107, 121) | 48.97 (33.28) | 50.32 (31.58)
  Week 52 (n=101, 119) | 50.17 (34.17) | 50.07 (31.62)

29. Secondary Outcome: Total Daily Long-Acting Insulin Dose Adjusted for Body Weight
Description: Total daily dose of long-acting insulin adjusted for body weight (units per kilogram [kg]). Long-acting insulin included Insulin NPH, Ultralente, and Insulin Glargine for both groups.
  Inhaled Insulin reported in mg/kg. Subcutaneous Insulin reported in units/kg.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 6, Week 9, Week 12, Week 18, Week 26, Week 39, Week 52
Population: Primary analysis set (PAS)
Measure: Mean (Standard Deviation); unit: mg/kg, units/kg
Groups:
- Inhaled Insulin (mg/kg): Inhaled insulin (Exubera®) with dose adjusted according to premeal blood glucose plus basal insulin.
- Subcutaneous Insulin (Units/kg): Subcutaneous insulin with dose adjusted according to premeal blood glucose plus basal insulin.
Arm/Group | Inhaled Insulin (mg/kg) | Subcutaneous Insulin (Units/kg)
Number analyzed (Participants) | 109 | 121
mg/kg, units/kg
  Baseline (n=105, 121) | 0.47 (0.25) | 0.52 (0.30)
  Week 1 (n=100, 112) | 0.47 (0.27) | 0.53 (0.31)
  Week 2 (n=103, 104) | 0.49 (0.29) | 0.52 (0.28)
  Week 3 (n=101, 113) | 0.49 (0.29) | 0.54 (0.31)
  Week 4 (n=99, 118) | 0.49 (0.27) | 0.54 (0.31)
  Week 6 (n=104, 121) | 0.52 (0.31) | 0.55 (0.32)
  Week 9 (n=99, 103) | 0.51 (0.31) | 0.54 (0.32)
  Week 12 (n=104, 117) | 0.52 (0.32) | 0.55 (0.32)
  Week 18 (n=108, 115) | 0.53 (0.33) | 0.55 (0.32)
  Week 26 (n=109, 120) | 0.52 (0.33) | 0.55 (0.32)
  Week 39 (n=105, 120) | 0.54 (0.37) | 0.56 (0.32)
  Week 52 (n=88, 108) | 0.53 (0.36) | 0.55 (0.31)

30. Secondary Outcome: Total Daily Short-Acting Insulin Dose (Unadjusted for Body Weight)
Description: Average Total Daily Insulin Dose: short-acting insulin (milligrams [mg]). Short-acting insulin (mg) for the Inhaled Insulin group was Inhaled Insulin. Short-acting insulin (unit) for the Subcutaneous Insulin group included Insulin Lispro, Insulin Aspart, and Regular Insulin.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 6, Week 9, Week 12, Week 18, Week 26, Week 39, Week 52
Population: Primary analysis set (PAS)
Measure: Mean (Standard Deviation); unit: mg, units
Arm/Group | Inhaled Insulin (mg) | Subcutaneous Insulin (Units)
Number analyzed (Participants) | 113 | 141
mg, units
  Baseline (n=109, 122) | 30.56 (22.69) | 30.74 (19.50)
  Week 1 (n=106, 118) | 11.03 (5.51) | 29.52 (19.95)
  Week 2 (n=108, 111) | 12.13 (6.03) | 31.24 (21.69)
  Week 3 (n=106, 116) | 12.96 (6.68) | 30.58 (20.70)
  Week 4 (n=106, 120) | 13.44 (6.82) | 31.87 (22.23)
  Week 6 (n=108, 122) | 14.04 (7.06) | 31.81 (21.94)
  Week 9 (n=106, 110) | 14.03 (7.76) | 31.55 (23.93)
  Week 12 (n=112, 122) | 14.42 (8.11) | 32.71 (23.70)
  Week 18 (n=112, 120) | 15.11 (8.68) | 33.49 (23.81)
  Week 26 (n=113, 122) | 15.95 (9.14) | 33.80 (24.37)
  Week 39 (n=109, 121) | 16.17 (10.25) | 33.12 (24.62)
  Week 52 (n= 103, 119) | 17.20 (10.95) | 33.04 (26.09)

31. Secondary Outcome: Total Daily Short-Acting Insulin Dose Adjusted for Body Weight
Description: Total Daily Short-Acting Insulin Dose adjusted for body weight (units divided by kg). Short-acting insulin (mg) for the Inhaled Insulin group was Inhaled Insulin. Short-acting insulin (unit) for the Subcutaneous Insulin group included Insulin Lispro, Insulin Aspart, and Regular Insulin.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 6, Week 9, Week 12, Week 18, Week 26, Week 39, Week 52
Population: Primary analysis set (PAS)
Measure: Mean (Standard Deviation); unit: mg/kg, units/kg
Arm/Group | Inhaled Insulin (mg/kg) | Subcutaneous Insulin (Units/kg)
Number analyzed (Participants) | 111 | 122
mg/kg, units/kg
  Baseline (n=109, 122) | 0.35 (0.25) | 0.36 (0.22)
  Week 1 (n=102, 113) | 0.12 (0.06) | 0.34 (0.23)
  Week 2 (n=104, 104) | 0.14 (0.07) | 0.36 (0.25)
  Week 3 (n=103, 112) | 0.15 (0.07) | 0.35 (0.23)
  Week 4 (n=101, 118) | 0.15 (0.07) | 0.37 (0.26)
  Week 6 (n=106, 121) | 0.16 (0.08) | 0.36 (0.24)
  Week 9 (n=101, 104) | 0.16 (0.09) | 0.36 (0.26)
  Week 12 (n=106, 117) | 0.16 (0.08) | 0.38 (0.26)
  Week 18 (n=110, 116) | 0.18 (0.10) | 0.37 (0.25)
  Week 26 (n=111, 121) | 0.19 (0.11) | 0.38 (0.27)
  Week 39 (n=107, 120) | 0.19 (0.12) | 0.38 (0.27)
  Week 52 (n=90, 108) | 0.19 (0.12) | 0.36 (0.29)

32. Secondary Outcome: Lipids: Median Change From Baseline to Last Observation
Description: Lipids: median changes (milligrams per deciliter [mg/dL]) from Baseline median to last observation in cholesterol (random), triglycerides (random), high density lipoprotein (HDL) cholesterol and low density lipoprotein (LDL) cholesterol. Normalized data was used in the computations. Last observation = last observation while on study drug or during the lag. Measures of dispersion for median changes in lipids were not determined.
Time Frame: Baseline to Last Observation
Population: Primary analysis set (PAS); median change from Baseline to last observation. Last observation was defined as last observation while on study drug or during the lag. Full range (-999 to 999) was not calculated.
Measure: Number; unit: mg/dL
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 110 | 121
mg/dL
  Cholesterol (random) (n=110, 121) | -0.5 (-0.5) [-999 to 999] | 0 (0) [-999 to 999]
  Triglycerides (random) (n=105, 121) | 9 (9) [-999 to 999] | -8 (-8) [-999 to 999]
  HDL Cholesterol (n=110, 121) | -3 (-3) [-999 to 999] | 1 (1) [-999 to 999]
  LDL Cholesterol (n=97, 110) | 0 (0) [-999 to 999] | 0 (0) [-999 to 999]

33. Secondary Outcome: Hypoglycemic Event Rates
Description: A Hypoglycemic event was identified by characteristic symptoms of hypoglycemia with no blood glucose check with prompt resolution with food intake, subcutaneous glucagon, or intravenouus glucose; characteristic symptoms with blood glucose of 59 milligrams per deciliter (mg/dL) (3.2 mmol/L) or less with blood glucose check; or any glucose measurement of 49 mg/dL (2.7 mmol/L) or less, with or without symptoms. Crude event rate = total events divided by subject months. Subject months = elapsed number of months a subject was in the study in each time interval.
Time Frame: 0 to 1 month to 11 to 12 months, and Overall
Population: Full analysis set (FAS)
Measure: Number; unit: events / subject-months
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 135 | 135
events / subject-months
  0 to 1 month (n=135, 135) | 2.99 | 2.48
  > 1 to 2 months (n=135, 135) | 2.52 | 2.34
  > 2 to 3 months (n=131, 134) | 2.12 | 1.84
  > 3 to 4 months (n=128, 134) | 1.84 | 1.61
  > 4 to 5 months (n=126, 134) | 1.94 | 1.69
  > 5 to 6 months (n=121, 131) | 1.51 | 1.84
  > 6 to 7 months (n=119, 131) | 1.50 | 1.67
  > 7 to 8 months (n=115, 129) | 1.45 | 1.26
  > 8 to 9 months (n=111, 129) | 1.62 | 1.26
  > 9 to 10 months (n=110, 129) | 1.26 | 1.55
  > 10 to 11 months (n=109, 125) | 1.12 | 1.37
  > 11 to 12 months (n=104, 123) | 1.18 | 1.23
  Overall (n=135, 135) | 1.79 | 1.68

34. Secondary Outcome: Severe Hypoglycemic Event Rates
Description: Severe hypoglycemic event = all 3 of the following criteria were met: subject unable to treat self, exhbited at least 1 neurological symptom (memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, suspected seizure, loss of consciousness); blood glucose measurement was ≤ 49 mg/dL, or not measured but clinical manifestations reversed by oral carbohydrates, subcutaneous glucagon, or i.v. glucose. Crude event rate = number of events divided by 100 subject-months. Subject months = elapsed number of months subject was in study in each time interval.
Time Frame: 0 to 1 month to 11 to 12 months, and Overall
Population: Full analysis set (FAS). Due the small number of events severe hypoglycemic event rates were assessed per 100 months.
Measure: Number; unit: Number of events/100 subject-months.
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 135 | 135
Number of events/100 subject-months.
  0 to 1 month (n=135, 135) | 2.91 | 1.48
  > 1 to 2 months (n=135, 135) | 5.22 | 1.49
  > 2 to 3 months (n=131, 134) | 4.64 | 2.99
  > 3 to 4 months (n=128, 134) | 0.78 | 2.24
  > 4 to 5 months (n=126, 134) | 4.05 | 1.51
  > 5 to 6 months (n=121, 131) | 3.33 | 2.29
  > 6 to 7 months (n=119, 131) | 0.00 | 0.77
  > 7 to 8 months (n=115, 129) | 0.89 | 2.33
  > 8 to 9 months (n=111, 129) | 5.42 | 1.55
  > 9 to 10 months (n=110, 129) | 0.91 | 3.18
  > 10 to 11 months (n=109, 125) | 1.88 | 2.41
  > 11 to 12 months (n=104, 123) | 3.95 | 3.10
  Overall (n=135, 135) | 2.89 | 2.13

35. Primary Outcome: Change From Baseline in Post-Bronchodilator Forced Expiratory Volume in One Second (FEV1)
Description: Change from Baseline at each visit in post-bronchodilator forced expiratory volume in one second (FEV1). FEV1 was measured in liters (L) 30 minutes following the administration of albuterol. Change from baseline: mean FEV1 (L) at observation minus baseline value.
Time Frame: Baseline through Week 52 Last Observation Carried Forward (LOCF)
Population: Full analysis set (FAS): all subjects who were randomized, had a baseline post-albuterol pulmonary function test (PFT) measurement, and had at least two post-baseline, post-albuterol PFT measurements. LOCF: last observation carried forward.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 141 | 139
liters
  Baseline (n=141, 139) | 2.559 (0.771) | 2.524 (0.742)
  Week 1 (n=123, 125) | -0.066 (0.150) | -0.027 (0.126)
  Week 2 (n=126, 115) | -0.056 (0.150) | -0.031 (0.128)
  Week 3 (n=131, 119) | -0.077 (0.185) | -0.030 (0.130)
  Week 4 (n=121, 129) | -0.074 (0.161) | -0.022 (0.155)
  Week 6 (n=130, 135) | -0.070 (0.248) | -0.025 (0.146)
  Week 12 (n=125, 129) | -0.053 (0.212) | -0.031 (0.182)
  Week 18 (n=124, 125) | -0.066 (0.226) | -0.040 (0.165)
  Week 26 (n=120, 128) | -0.056 (0.175) | -0.038 (0.184)
  Week 39 (n=107, 124) | -0.088 (0.191) | -0.039 (0.194)
  Week 52 (n=106, 112) | -0.131 (0.259) | -0.059 (0.234)
  Week 52 LOCF (n=141, 139) | -0.113 (0.261) | -0.062 (0.225)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.039, 90% CI [-0.079 to -0.000], Standard Error of Mean 0.024
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.029, 90% CI [-0.068 to 0.010], Standard Error of Mean 0.024
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.045, 90% CI [-0.084 to -0.006], Standard Error of Mean 0.024
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.046, 90% CI [-0.085 to -0.007], Standard Error of Mean 0.024
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.046, 90% CI [-0.085 to -0.007], Standard Error of Mean 0.024
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.023, 90% CI [-0.063 to 0.017], Standard Error of Mean 0.024
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.021, 90% CI [-0.062 to 0.020], Standard Error of Mean 0.025
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.014, 90% CI [-0.055 to 0.027], Standard Error of Mean 0.025
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.042, 90% CI [-0.085 to 0.000], Standard Error of Mean 0.026
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.065, 90% CI [-0.109 to -0.022], Standard Error of Mean 0.027
Statistical Analysis 11: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52 Last Observation Carried Forward (LOCF; Inhaled Insulin - Subcutaneous Insulin. Adjusted (primary analysis model) includes terms of Treatment, Week, Baseline pulmonary function test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.050, 90% CI [-0.097 to -0.003], Standard Error of Mean 0.028

36. Primary Outcome: Change From Baseline in Post-Bronchodilator Carbon Monoxide Diffusing Capacity (DLco)
Description: Carbon Monoxide Diffusing Capacity (DLco) measured in milliters/minutes/millimeters of mercury (mL/min/mmHg) 30 minutes following the administration of albuterol. Change from Baseline: mean DLco (mL/min/mmHg) at observation minus baseline value.
Time Frame: as for outcome 3
Population: Full analysis set (FAS); LOCF: last observation carried forward.
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 141 | 139
mL/min/mmHg
  Baseline (n=141, 139) | 23.023 (5.914) | 22.883 (6.079)
  Week 1 (n=122, 124) | -0.574 (1.392) | -0.333 (1.405)
  Week 2 (n=126, 112) | -0.777 (1.631) | -0.481 (1.290)
  Week 3 (n=129, 118) | -0.811 (1.244) | -0.506 (1.388)
  Week 4 (n=120, 128) | -1.075 (1.425) | -0.576 (1.397)
  Week 6 (n=129, 135) | -1.017 (1.633) | -0.602 (1.488)
  Week 12 (n=125, 125) | -0.961 (1.738) | -0.477 (1.588)
  Week 18 (n=124, 123) | -1.024 (1.774) | -0.549 (1.601)
  Week 26 (n=119, 127) | -0.849 (1.914) | -0.477 (1.706)
  Week 39 (n=107, 123) | -1.016 (1.649) | -0.395 (1.767)
  Week 52 (n=105, 110) | -1.483 (1.944) | -0.798 (1.967)
  Week 52 LOCF (n=141, 139) | -1.426 (1.856) | -0.682 (1.958)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.279, 90% CI [-0.606 to 0.048], Standard Error of Mean 0.199
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.336, 90% CI [-0.661 to -0.011], Standard Error of Mean 0.198
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.384, 90% CI [-0.707 to -0.061], Standard Error of Mean 0.196
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.516, 90% CI [-0.842 to -0.191], Standard Error of Mean 0.198
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.474, 90% CI [-0.797 to -0.152], Standard Error of Mean 0.196
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.533, 90% CI [-0.866 to -0.200], Standard Error of Mean 0.202
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.509, 90% CI [-0.845 to -0.174], Standard Error of Mean 0.204
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.412, 90% CI [-0.749 to -0.076], Standard Error of Mean 0.204
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.707, 90% CI [-1.056 to -0.358], Standard Error of Mean 0.212
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.680, 90% CI [-1.040 to -0.320], Standard Error of Mean 0.219
Statistical Analysis 11: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Week 52 Last Observation Carried Forward (LOCF); Inhaled Insulin - Subcutaneous Insulin. Adjusted (primary analysis model) includes terms of Treatment, Week, Baseline pulmonary function test (PFT), Center, Age, Sex, Baseline Height, Type of Diabetes, and Controller Medications Use on Day of Randomization; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.765, 90% CI [-1.116 to -0.415], Standard Error of Mean 0.212

ADVERSE EVENTS:
Description: Adverse events for this study are reported using MedDRA in these Basic Results, but are reported using COSTART in the Clinical Study Report and PhRMA Web Synopsis for consistency with earlier studies. Consequently, subtle differences may be observed.
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Serious Adverse Events (participants affected / at risk) | 21/146 | 13/141
Other Adverse Events (participants affected / at risk) | 140/146 | 136/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Insulin (N=146) | Subcutaneous Insulin (N=141)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 2 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Insulin (N=146) | Subcutaneous Insulin (N=141)
Conjunctivitis (Eye disorders) | 3 | 9
Constipation (Gastrointestinal disorders) | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 10 | 6
Nausea (Gastrointestinal disorders) | 12 | 8
Vomiting (Gastrointestinal disorders) | 8 | 5
Chest pain (General disorders) | 8 | 7
Fatigue (General disorders) | 9 | 7
Oedema peripheral (General disorders) | 11 | 14
Seasonal allergy (Immune system disorders) | 3 | 7
Bronchitis (Infections and infestations) | 24 | 18
Gastroenteritis (Infections and infestations) | 8 | 7
Gastroenteritis viral (Infections and infestations) | 5 | 7
Influenza (Infections and infestations) | 20 | 25
Nasopharyngitis (Infections and infestations) | 29 | 26
Sinusitis (Infections and infestations) | 14 | 21
Upper respiratory tract infection (Infections and infestations) | 44 | 39
Urinary tract infection (Infections and infestations) | 18 | 20
Hypoglycaemia (Metabolism and nutrition disorders) | 109 | 120
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 15
Tendonitis (Musculoskeletal and connective tissue disorders) | 4 | 8
Dizziness (Nervous system disorders) | 11 | 10
Headache (Nervous system disorders) | 14 | 14
Neuropathy peripheral (Nervous system disorders) | 2 | 7
Tremor (Nervous system disorders) | 8 | 17
Depression (Psychiatric disorders) | 11 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 53 | 63
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 13

LIMITATIONS AND CAVEATS:
Data for some secondary endpoints were not tabulated or analyzed for this study and some concomitant medication data were not accurately recorded and tabulated due to lack of resources resulting from scaling down of Exubera® development.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.